CLINICAL TRIAL: NCT04278443
Title: A Single Site Prospective Descriptive Study on the Effect of Brachytherapy Monotherapy for Prostate Cancer on Male Fertility
Brief Title: Fertility After Prostate Brachytherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: BXTAccelyon Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: RD2016-50
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and semen samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low dose rate brachytherapy: 20 patients receiving low dose rate brachytherapy
- High dose rate brachytherapy: 20 patients receiving high dose rate brachytherapy.

SUMMARY:
Although brachytherapy toxicity data on erectile dysfunction, urethral dysfunction and bladder and bowel impact has been collected for a number of years, there is limited information on its effect on male fertility. This study aims to investigate the effect of brachytherapy on fertility

DETAILED DESCRIPTION:
Brachytherapy is a commonly employed technique in the treatment of all prostate cancer risk groups. It delivers a high radiation localised to the prostate gland. The effects of this on fertility have not been systematically studied. An increasing number of younger men for whom fertility is an issue are being diagnosed with prostate cancer and may be offered brachytherapy amongst their treatment choices. This study therefore addresses this issue with a systematic evaluation of sperm count and quality before and after both high dose rate and low dose rate brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 years or older
* Receiving brachytherapy monotherapy; High or Low dose rate
* Ability to ejaculate
* Able to provide written informed consent

Exclusion Criteria:

* History of infertility or vasectomy
* Previous chemotherapy or pelvic radiotherapy
* Prior use of androgen deprivation therapy
* 5 alpha-reductase inhibitors within the last 4 months
* Alpha blockers within 7 days of semen collection

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Study on male fertility, thus only male participants are eligible
Study Population: Men undergoing brachytherapy for prostate cancer
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-02-24 (Actual); Primary Completion 2021-08-05 (Estimated); Study Completion 2021-08-05 (Estimated)

PRIMARY OUTCOMES:
To define effect of prostate brachytherapy on male fertility. | 12 months
  measure by sequential sperm counts

CONTACTS AND LOCATIONS:
Locations (1):
- East and North Hertfordshire NHS Trust, Northwood, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided